CLINICAL TRIAL: NCT01331434
Title: A Single Dose, 2-Period, 2-Treatment, 2-Way Bioequivalency Study of Exemestane 25 mg Tablets Under Fed Conditions
Brief Title: Bioequivalency Study of Exemestane 25 mg Tablet Under Fed Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roxane Laboratories (Industry)
Responsible Party: Elizabeth Ernst, Executive Director, Drug Regulatory Affairs and Medical Affairs, Roxane Laboratories, Inc.
Organization: West-Ward Pharmaceutical (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: EXEM-02
Record Dates: First submitted 2011-04-06; First posted 2011-04-08 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — exemestane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: exemestane — 25 mg tablet
  Other Names: AROMASIN

SUMMARY:
The objective of this study was to prove the bioequivalence of Exemestane 25 mg tablet under fed conditions.

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant abnormal findings on the physical examination, medical history, or clinical laboratory results during screening

Exclusion Criteria:

* Positive test for HIV, Hepatitis B, or Hepatitis C.
* Treatment with known enzyme altering drugs.
* History of allergic or adverse response to exemestane or any comparable or similar product.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2004-10; Primary Completion 2004-10 (Actual); Study Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
bioequivalence determined by statistical comparison Cmax | 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Dennis N Morrison, D.O., Principal Investigator — Bio-Kinetic Clinical Applications, Inc.
Locations (1):
- Bio-Kinetic Clinical Applications, Inc., Springfield, Missouri, United States